CLINICAL TRIAL: NCT07125950
Title: A Phase 2 Trial of SHR2554 Combined With Endocrine Therapy in Advanced Breast Cancer
Brief Title: SHR2554 Combined With Endocrine Therapy in Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief physician, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-IIT-SHR2554-ET
Record Dates: First submitted 2025-08-06; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1 (Experimental): SHR2554+HRS-8080
  Interventions: Drug: SHR2554; Drug: HRS-8080
- Arm2 (Experimental): SHR2554+HRS-1358
  Interventions: Drug: SHR2554; Drug: HRS-1358

INTERVENTIONS:
Drug: SHR2554 — SHR2554
Drug: HRS-8080 — HRS-8080
  Arms: Arm1
Drug: HRS-1358 — HRS-1358
  Arms: Arm2

SUMMARY:
Our study is aimed to evaluate the safety and preliminary of all-oral regimen SHR2554 combined with HRS-8080 or HRS-1358 in advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years old (including boundary values), patients with advanced or metastatic breast cancer;
* ECOG PS Score: 0~1;
* Based on RECIST v1.1, at least one measurable lesion;
* Patients must have a life expectancy ≥ 3 months;
* Adequate organ function and marrow function (no corrective treatment within 14 days before first dose);
* Women of childbearing potential (WOCBP) should agree to use an effective method of contraception and no lactation from the initiation of screening to 7 months after the last dose of study therapy; WOCBP should have a negative serum pregnancy result within 7 days before the first dose of study therapy; if unneutered male subjects (including using other sterilization except bilateral orchidectomy [e.g. vasectomy]) are willing to have sexual behaviour with WOCBP, one kind of contraception must be used to prevent the pregnancy of his partner from the date of enrolment to 7 months after the last dose of study therapy);
* Willing and able to provide written informed consent and comply with the requirements and restrictions in the protocol.

Exclusion Criteria:

* Has received or been receiving ADC therapy;
* Active brain metastasis (without medical control or having clinical symptoms), carcinomatous meningitis or spinal compression;
* Existence of third space fluid (e.g. massive ascites, pleural effusion) which is not well controlled by effective methods, e.g. drainage, evaluated by investigators;
* Other malignancy within prior 2 years with no necessary treatment (except hormone replacement treatment) for at least recent 2 years, except: curatively treated in situ cancer of the cervix, skin basal cell carcinoma, skin squamous cell carcinoma or papillary thyroid carcinoma;
* Has received antitumor surgery, radiotherapy, chemotherapy, targeted therapy or immunological therapy within 2 weeks or 5-fold half-life of drugs (whichever is shorter) before first dose of study therapy; has received antitumor endocrine therapy within one week before first dose of study therapy;
* Adverse events caused by prior antitumor therapy have not recovered to ≤grade 1 per NCI-CTCAE v5.0 (except alopecia and tolerable, chronic grade 2 toxicity determined by investigator);
* Use of other antitumor systemic treatment during the study;
* Has received CYP3A4 median or potent inhibitors within 2 weeks before the first dose, or CYP3A4 median or potent inducers within 4 weeks before the first dose, or been receiving known CYP3A5 median or potent inhibitors or inducers;
* Hypersensitivity to study therapy or any of its excipients;
* Uncontrolled chronic, systemic complicating disease evaluated by investigators (e.g. severe, chronic pulmonary, hepatic, renal or heart disease);
* Known history of immunodeficiency, including HIV-positive, other acquired or innate immunodeficient disease, or known history of organ transplantation, or known history of allogenic haemopoietic stem cell transplantation;
* Has active hepatitis B (HBsAg-positive and HBV DNA≥500 IU/mL), hepatitis C (positive for HCV antibody and HCV RNA above ULN) and hepatic cirrhosis;
* Has an active infection requiring antibiotics, antiviral or antifungal treatment, or pyrexia >38.5℃ of unknown origin during the screening period before first dose of study therapy (patients with pyrexia due to cancer could be enrolled determined by investigator);
* Known clinically severe cardiac-cerebral vascular disease, including: (1) congestive heart failure (NYHA Class >2); (2) unstable angina pectoris; (3) myocardial infarction over the past year; (4) any supraventricular or ventricular arrhythmia needed to treat or intervene; ECG abnormality of clinical significance evaluated by investigators; existence of arterial/venous thrombotic event within 6 months before first dose, or cerebrovascular accidents, or transient ischemic attack;
* Inability to take oral medication (e.g., unable to swallow, intestinal obstruction), or any active gastrointestinal disease or other condition resulting in inability to drug absorption, distribution, metabolism or excretion (e.g., active gastroenteritis, chronic diarrhoea, intestinal syndrome, or upper gastrointestinal surgery, including gastrectomy);
* Other conditions that might influence the study and analysis of results in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator | At baseline, at the time point of every 8 weeks within first 24 weeks, thereafter every 12 weeks
  ORR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response) or PR (partial response) per RECIST v1.1.

SECONDARY OUTCOMES:
CBR by investigator | At baseline, at the time point of every 8 weeks within first 24 weeks, thereafter every 12 weeks
  CBR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response), PR (partial response) or SD (stable disease)≥6 months per RECIST v1.1.
DoR | up to 3 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
PFS | up to 3 years
  PFS is the time from the date of first dose until the date of objective radiographic disease progression or death (by any cause in the absence of progression).
OS | up to 3 years
  OS is the time from the date of first dose until the date of death by any cause.
Safety (Proportion of AEs) | from time of informed consent provided to 30 days after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experienced an adverse event and discontinued study drug due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Chief physician, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No